CLINICAL TRIAL: NCT01803451
Title: The Role of Glucagon Like Peptide-1 in Glucose Metabolism and Weight Loss Following Gastric Bypass Surgery
Brief Title: Glucagon-like Peptide 1, Glucose Metabolism and Gastric Bypass
Acronym: GLP-1
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: HSC20180070H; DK083554 (Other: NIDDK)
Record Dates: First submitted 2013-02-20; First posted 2013-03-04 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Post-bariatric Surgery
Keywords: gastric bypass; glucose metabolism; hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — exendin (9-39)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hyperglycemic clamp-Meal tolerance test (Experimental): these studies are to evaluate the effect of exendin-9 on insulin secretion before and after meal ingestion in patients after bariatric surgeries compared to non-surgical controls
  Interventions: Drug: exendin-(9-39)
- Labeled meal tolerance test (Experimental): The effect of GLP-1 receptor blockade on glucose tolerance and glucose kinetics are evaluated in the group patients with bariatric surgery vs. nonsurgical using exendin-9-39 infusion during one of the the 2-day dual tracer studies of meal tolerance test
  Interventions: Drug: exendin -(9-39)

INTERVENTIONS:
Drug: exendin-(9-39) — hyperglycemic clamp-meal tolerance test is designed to assess insulin secretion before and after meal ingestion
  Other Names: no other name for exendin-(9-39)
  Arms: hyperglycemic clamp-Meal tolerance test
Drug: exendin -(9-39) — 2-day meal tolerance tests with labeled oral and IV glucose using exendin-(9-39) infusion are designed to evaluate the role of GLP-1 signaling on glucose tolerance and glucose kinetics.
  Other Names: no other name for exendin-(9-39)
  Arms: Labeled meal tolerance test

SUMMARY:
The overall goal of this project is to understand the mechanisms by which gastric bypass surgery improves glucose metabolism.

The central hypothesis guiding this project is that the reconfiguration of intestinal transit with the Roux-en-Y will increase the release of insulinotropic GI hormones, termed incretins that improve insulin secretion and glucose metabolism. The study is divided into three specific aims.

1. To determine the role of incretin hormones on insulin secretion in patients with gastric bypass surgery using intravenous-oral hyperglycemic clamp.
2. To compare incretin effect and glucose tolerance among patient who suffer from hypoglycemia after RYGB and asymptomatic surgical and non-surgical individuals.
3. To quantify the contribution of GLP-1 to incretin effect enhancement following surgery.

DETAILED DESCRIPTION:
The overall goal of this project is to understand the mechanisms by which gastric bypass surgery improves glucose metabolism.

The central hypothesis guiding this project is that the reconfiguration of intestinal transit with the Roux-en-Y will increase the release of insulinotropic GI hormones, termed incretins that improve insulin secretion and glucose metabolism. The study is divided into three specific aims.

1. To determine the role of incretin hormones on insulin secretion in patients with gastric bypass surgery using intravenous-oral hyperglycemic clamp.
2. To compare incretin effect and glucose tolerance among patient who suffer from hypoglycemia after RYGB and asymptomatic surgical and non-surgical individuals.
3. To quantify the contribution of GLP-1 to incretin effect enhancement following surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* healthy control without diabetes or active organ disease
* Individuals with bariatric surgery
* recurrent hypoglycemia post gastric bypass

Exclusion Criteria:

* pregnancy
* significant anemia
* diabetes currently unless pre-op for bariatric surgery procedure
* GI obstruction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-11; Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
The investigator measure glucose, islet and GI hormonal levels in response to meal ingestion as a composite measure and the percentage of contribution of GLP-1 contribution to postprandial insulin levels will also be calculated | up to 1 year (10 sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Marzieh Salehi, MD,MS, Principal Investigator — Marzieh Salehi
Locations (2):
- United States (2):
  - Texas Diabetes Institute - University Health System, San Antonio, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas

REFERENCES:
- [Derived] Salehi M, Gastaldelli A, D'Alessio DA. Blockade of glucagon-like peptide 1 receptor corrects postprandial hypoglycemia after gastric bypass. Gastroenterology. 2014 Mar;146(3):669-680.e2. doi: 10.1053/j.gastro.2013.11.044. Epub 2013 Dec 4. PMID 24315990